CLINICAL TRIAL: NCT06674707
Title: Effects of Agility Training With and Without Foot Mobilization On Pain, Balance and Functional Performance In Patellofemoral Pain Syndrome.
Brief Title: Effects of Agility Training With and Without Foot Mobilization In Patellofemoral Pain Syndrome.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/24/0131
Record Dates: First submitted 2024-11-03; First posted 2024-11-05 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-11

CONDITIONS: Patellofemoral Pain Syndrome
Keywords: Balance; Functional Performance; Flat foot; Kujala function scale; Patellofemoral pain syndrome; Pain
MeSH Terms: conditions — Patellofemoral Pain Syndrome; Flatfoot; Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Agility Training with Foot Mobilization (Experimental): Agility Training with Foot Mobilization along with simple conventional treatment
  Interventions: Other: Agility Training with Foot mobilization.
- Agility Training without Foot Mobilization. (Active Comparator): Agility training without foot mobilization along with simple conventional treatment.
  Interventions: Other: Agility Training without Foot mobilization

INTERVENTIONS:
Other: Agility Training with Foot mobilization. — Agility training with foot mobilization with the frequency of 3 sets of 10 repetitions thrice per week for a total six weeks. Pre and post intervention values will be taken on 1st day and after six weeks. Agility training includes side stepping, braiding activities, and front and back crossover steps during forward ambulation, shuttle walking, multiple changes in direction during walking on therapist command. TJM is a grade III Maitland technique and is applied with a high amplitude from the end range and 1s of vibration in the middle range of the joint through a linear motion to where tissue resistance is felt in the prone position, the patient is supported by a towel placed under the foot. Two sets of 5 min total were performed for 6weeks.
  Other Names: Simple conventional Treatment
  Arms: Agility Training with Foot Mobilization
Other: Agility Training without Foot mobilization — Agility training includes side stepping, braiding activities, and front and back crossover steps during forward ambulation, shuttle walking, multiple changes in direction during walking on therapist command. Comprising of Hot pack and TENS for 10 minutes and Ultrasound for 5 minutes . Comprising of conventional exercises were given for 3 sessions per week for 6 weeks. It includes semi squat, quadriceps isometric, terminal knee extension with elastic band, terminal knee extension in supine position, and adductor squeeze in crook lying (squeeze the ball).
  Other Names: Simple Conventional Treatment
  Arms: Agility Training without Foot Mobilization.

SUMMARY:
Patellofemoral pain syndrome (PFPS) is referred to as peripatellar or retro-patellar pain, which is characterized by alterations in the physical and biomechanical features of the patellofemoral joint. Risk factors for PFPS include: anatomic anomalies, mal-alignment and altered biomechanics of the lower extremity, muscle dysfunction, patellar hypermobility, poor quadriceps, or iliotibial band flexibility, surgery, tight lateral structures, training errors or overuse and trauma. The aim of this study is to compare the effects of foot mobilization with and without agility training on pain, balance and functional performance in patellofemoral pain syndrome.

DETAILED DESCRIPTION:
A Randomized Clinical Trial will be conducted at Riphah Clinic Lahore, Al Rehman Hospital, through convenient purposive sampling technique on 42 patients which will be allocated through using simple randomization into Group A and Group B. Group A will be treated with agility training and foot mobilization in patellofemoral pain syndrome and Group B will be treated with agility training without foot mobilization in patellofemoral pain syndrome thrice a week for 6 weeks. Outcome measures will be conducted through pain (NPRS), Kujala patellofemoral pain scale, Y balance test and Navicular droop test before and after 6 weeks. Data will be analyzed using SPSS software version 25.

ELIGIBILITY:
Inclusion Criteria:

Clinical signs of patellofemoral pain syndrome such as retro patellar pain, crepitation, and pain with patellar grinding more than 6 months.

* Both genders of 20-40 years of age.
* Presence of pain on step down from a 25 step or double leg squat and sitting with knee bent greater than 15 min.
* Pain more than 4 on NPRS scale.
* Individual with anterior left/right asymmetries greater than 4 cm on Y balance test
* Excessive calcaneal eversion measured at 6° in the relaxed posture(6).

Exclusion Criteria:

* History of ligament and meniscal injury.
* History of lower limb fractures.
* History of post-surgical condition of lower limb
* History of systemic, connective tissue or neurologic condition

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 42 (Estimated)
Dates: Start 2024-01-04 (Actual); Primary Completion 2025-01-07 (Estimated); Study Completion 2025-01-07 (Estimated)

PRIMARY OUTCOMES:
Numeric Pain Rating Scale (NPRS): | 6 weeks
  The outcome was the 11-point NPRS to measure pain intensity. The NPRS defines pain intensity from 0 to 10 points, with 0 and 10 points indicating no pain and the most severe pain respectively. The reported test-retest reliability (intraclass correlation coefficient [ICC]) was 0.76, demonstrating it to be a good indicator of pain intensity.
Kujala Patellofemoral Pain Scale | 6 weeks
  Anterior knee pain scale is frequently referred as Kujala scale. It's a 13 item questionnaire including different items on pain related to function and activities. The items assessed in the questionnaire are patellar subluxation, claudication, pain, walking, climbing stairs and prolonged sitting with the knees flexed. It has a score from 0 to 100 points, where 100 means without pain and functional limitations and 0 means constant pain and various functional limitations.
Y Balance Test | 6 weeks
  The YBT assesses the balance by challenging his postural control system in 3 (anterior, posteromedial, and posterolateral) of the 8 SEBT (star excursion balance test) directions and has been advocated as a method for assessing dynamic balance (requires strength, flexibility and proprioception). The Y balance score was calculated by dividing the sum of the maximum reach distance in the anterior (A), posteromedial (PM), and posterolateral (PL) directions by 3 times the limb length (LL) of the individual, then multiplied by 100.
Navicular Droop Test | 6 weeks
  Position the patient in standing so there is full weight-bearing through the lower extremity and ensure the foot is in the subtalar joint neutral position ("talar head congruent"). Mark the most prominent part of the navicular tuberosity and measure its distance from the supporting surface floor or step. Ask the patient to relax and then measure the amount of sagittal plane excursion of the navicular with a ruler. Alternatively, the test can also be performed in reverse, measuring from relaxed position up to talar neutral in standing postion. Many clinicians also choose to perform this test by marking the start and end position of the navicular on an index card placed along the inside of the foot and then measure the change with a ruler. The ICC2,1 values in the sitting and standing positions were 0.93 and 0.95, respectively, indicating significantly high inter-rater reliability.

CONTACTS AND LOCATIONS:
Overall Officials: Ali Raza, MS-OMPT, Principal Investigator — Riphah International University
Locations (1):
- Al- Rehman Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Luza LP, Luza M, Santos GM. Patellofemoral Pain Syndrome Modifies the Movement of the Rearfoot, but It Does Not Alter Plantar Pressure Distribution. Rev Bras Ortop (Sao Paulo). 2020 Aug;55(4):419-425. doi: 10.1055/s-0039-1698802. Epub 2019 Dec 13. PMID 32904777
- [Background] Gomez Carrion A, de Los Angeles Atin Arratibel M, Morales Lozano MR, Martinez Sebastian C, de la Cruz Torres B, Sanchez-Gomez R. Kinematic Effect on the Navicular Bone with the Use of Rearfoot Varus Wedge. Sensors (Basel). 2022 Jan 21;22(3):815. doi: 10.3390/s22030815. PMID 35161560
- [Background] Rasti E, Rojhani-Shirazi Z, Ebrahimi N, Sobhan MR. Effects of whole body vibration with exercise therapy versus exercise therapy alone on flexibility, vertical jump height, agility and pain in athletes with patellofemoral pain: a randomized clinical trial. BMC Musculoskelet Disord. 2020 Oct 26;21(1):705. doi: 10.1186/s12891-020-03732-1. PMID 33106162
- [Background] Adhama AI, Akindele MO, Ibrahim AA. Effects of variable frequencies of kinesthesia, balance and agility exercise program in adults with knee osteoarthritis: study protocol for a randomized controlled trial. Trials. 2021 Jul 21;22(1):470. doi: 10.1186/s13063-021-05386-3. PMID 34289884
- [Background] Shakouri A, Kamali F, Mohamadi M, Nouhi E. Lumbopelvic manipulation alone versus combined with dry needling in physically active patients with patellofemoral pain syndrome: A randomized clinical trial. J Bodyw Mov Ther. 2024 Jan;37:220-225. doi: 10.1016/j.jbmt.2023.11.024. Epub 2023 Nov 25. PMID 38432809
- [Background] da Silva Boitrago MV, de Mello NN, Barin FR, Junior PL, de Souza Borges JH, Oliveira M. Effects of proprioceptive exercises and strengthening on pain and functionality for patellofemoral pain syndrome in women: A randomized controlled trial. J Clin Orthop Trauma. 2021 Apr 19;18:94-99. doi: 10.1016/j.jcot.2021.04.017. eCollection 2021 Jul. PMID 33996453
- [Background] Clifford AM, Dillon S, Hartigan K, O'Leary H, Constantinou M. The effects of McConnell patellofemoral joint and tibial internal rotation limitation taping techniques in people with Patellofemoral pain syndrome. Gait Posture. 2020 Oct;82:266-272. doi: 10.1016/j.gaitpost.2020.09.010. Epub 2020 Sep 15. PMID 32987346